CLINICAL TRIAL: NCT07397065
Title: Moni-Patc Temperature Monitoring Patch System Clinical Accuracy Validation
Brief Title: Clinical Accuracy Validation of the Moni-Patc Temperature Monitoring Patch During Surgery (Compared With Esophageal and Bladder Temperature)
Acronym: Moni-Patch OR
Status: Not yet recruiting | Type: Observational
Sponsor: Murata Vios, Inc. (Industry)
Collaborators: University of Minnesota (Other)
Responsible Party: Sponsor
Other Study IDs: MM-MPS2-0001
Record Dates: First submitted 2026-01-28; First posted 2026-02-09 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Temperature Monitoring; Intraoperative

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

INTERVENTIONS:
Device: Moni-Patc Temperature Monitoring Patch System — A non-sterile, non-invasive temperature monitoring system applied to the neck; Bluetooth 5.0 transmission to a receiver; continuous core temperature estimation using dual heat-flux/thermistor-based algorithm; conforms to ISO 80601-2-56 (25-42 °C).
  Other Names: MP-P20U Sensor; MP-D20U Receiver; MP-S20U Disposable Strips; MP-E20U Extension Cable

SUMMARY:
Moni-Patc Temperature Monitoring Patch System, a non-invasive, continuous temperature monitoring device designed to estimate core body temperature by applying a Sensor to the neck.This clinical accuracy validation study aims to verify the accuracy and repeatability of the Moni-Patch compared with an FDA-cleared continuous esophageal and bladder temperature monitoring device used as the clinical reference.Main ObjectivesTo verify that the Moni-Patch and the reference device(esophageal and bladder) demonstrate acceptable agreement, as defined by Bland-Altman Analyses (bias within ±0.4°C and limits of agreement between -1.0°C and 1.0°C).To verify the consistency and repeatability of temperature measurements obtained from the Moni-Patch during continuous monitoring.

DETAILED DESCRIPTION:
This single-center, open-label accuracy validation compares continuous core temperature measured by the Moni-Patch applied on the neck with esophageal (T_eso) and bladder (T_bld) temperatures during elective surgeries under general anesthesia. Approximately 30 adult participants will be monitored for ≥60 minutes intraoperatively. Agreement will be assessed using Bland-Altman methods (bias and 95% limits of agreement). The device is non-invasive and Bluetooth-enabled; readings are captured via the receiver and routed to the OR multi-parameter monitor and EMR. Safety monitoring focuses on device-related skin reactions and device deficiencies; no changes to anesthetic care are mandated by the protocol.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years
2. Subject is undergoing an elective surgical procedure expected to require at least 60min of general anesthesia and during which routine esophageal (Teso) and bladder (Tbld) temperature monitoring is expected.
3. Subjects are expected to remain hospitalized at least overnight after surgery.
4. Subject specifically agrees to temperature Sensor placement on the neck prior to surgery.
5. Must be able to attach the Sensor away from the operative field (neck) with uninterrupted wireless connection between the Sensor and the Receiver (as close as possible).
6. Use environment must meet both of the following parameters:

   1. Temperature 15-40⁰ C/59-104⁰ F
   2. Humidity 30-75% RH (non-condensing)
7. For non-English speaking subjects, a translator must be present at the time of consent.

Exclusion Criteria:

1. Subjects unable to provide their own consent. Consent from family or LOR is not acceptable.
2. Subjects undergoing surgical procedures who have conditions of the esophagus or bladder that contraindicate placement of these monitoring probes/sensor.
3. Subjects whose surgery does not involve the monitoring of esophageal or bladder temperature.
4. Subjects undergoing surgery that prohibits placement of an esophageal temperature monitoring probe/sensor (e.g. neck surgery).
5. Subjects with medical conditions such as inflammation, scratches, redness, rash at the Sensor placement site.
6. Subjects for whom the sensor cannot be securely adhered to the skin without floating or detaching, or accurately positioned over the carotid artery.
7. Not for use in MRI or CT facilities.
8. Use environment does not meet one or more parameters.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population consists of adult patients aged 18 years and older who are undergoing elective surgical procedures under general anesthesia in the operating room. Eligible participants are those for whom continuous esophageal and bladder temperature monitoring is clinically indicated as part of routine perioperative care and who are expected to remain hospitalized overnight following surgery.
  Participants will have the Moni-Patch Temperature Monitoring Patch System applied to the neck for continuous, non-invasive temperature monitoring during surgery. The study population will include a range of body mass index (BMI) categories to support evaluation of device performance across different body habitus. Subjects must be able to provide informed consent and meet environmental and clinical conditions required for use of the study device.
Sampling Method: Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2026-02-06 (Estimated); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Agreement Between Moni-Patch™ Temperature Monitoring Patch System and Esophageal (Teso) and Bladder (Tbld) Core Temperature Measurements | Continuous intra-operative monitoring for ≥60 minutes, beginning after ≥30 minutes of Moni-Patch sensor acclimation prior to operating room entry.
  This outcome assesses agreement between the Moni-Patch™ Temperature Monitoring Patch System and clinical reference core temperature measurements obtained using FDA-cleared esophageal temperature probes (Teso) and FDA-cleared bladder temperature probes (Tbld) during general anesthesia.
  Paired temperature values are collected simultaneously from:
  Moni-Patch™ Sensor (neck placement) Esophageal core temperature probe (Teso) Bladder core temperature probe (Tbld)
  Agreement is evaluated using Bland-Altman analysis, including:
  Mean temperature difference (bias; °C) 95% limits of agreement (LOA; °C)
  Name of Measurement: Core temperature difference (Moni-Patch - Teso; Moni-Patch - Tbld)
  Measurement Tools:
  Moni-Patch™ Temperature Monitoring Patch System FDA-cleared esophageal core temperature monitor (Teso) FDA-cleared bladder core temperature monitor (Tbld) Unit of Measure: Degrees Celsius (°C)

IPD SHARING:
Plan to Share IPD: No
De-identified device signal data may be shared upon reasonable request after publication, subject to data use agreement; no PHI will be shared.